CLINICAL TRIAL: NCT02811172
Title: Behavior of Biomarkers During Pregnancy and Lactation Through a Biological Multi-paradigm Model: BECOME Study Protocol
Acronym: BECOME
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor, Universidad de Granada
Other Study IDs: SPID201600X080546IV0
Record Dates: First submitted 2016-05-17; First posted 2016-06-23 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy; Gestational Diabetes; Hypertension; Obesity
Keywords: Biological multi-paradigm model; Biomarkers; Triglycerides; Cholesterol; Prolactin; Glucose
MeSH Terms: conditions — Diabetes, Gestational; Hypertension; Obesity | interventions — Lactation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Triglycerides; Cholesterol; Prolactin; Glucose; Human Milk.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy pregnant women: Healthy pregnant women
  Interventions: Other: BEhavior of biomarkers during pregnanCy and lactatiOn
- Risk pregnant women: Hypertensive, obese and diabetic women
  Interventions: Other: BEhavior of biomarkers during pregnanCy and lactatiOn

INTERVENTIONS:
Other: BEhavior of biomarkers during pregnanCy and lactatiOn

SUMMARY:
Background Despite of advances in research, at the moment, various points related to the physiology of gestation and the etiology of severe diseases that can be developed in the course of it remain unknown. One of those aspects is the behavior of biomarkers (triglycerides, prolactin, glucose and cholesterol) during pregnancy, which experience a gradual increase in their levels until they reach the peak of hypertriglyceridemia, a few days before delivery. Several studies have reported that biomarkers experience a higher elevation in diabetic and obese pregnant women and in those women who suffer preeclampsia. The description of their behavior in different population of pregnant women (healthy women and women at risk) would identify the relation of these with some of the alterations that occurs more frequently during pregnancy.

Objective The aim of this study is to develop a multi-paradigm biological model of systems to determine triglyceride, prolactin, glucose and cholesterol levels during pregnancy and its relation with lactogenesis in healthy and risk pregnant women.

Methods A prospective cohort study will take place with women during pregnancy and lactation. Participating women will be divided into two groups. One group will be integrated by healthy women and the other group by pregnant women with a risk medical history. The personal, family and a detailed medical history will be collected in each group. A study of all the variables which influence the level of the mentioned biomarkers (triglycerides, cholesterol, glucose and prolactin) will be done.

The universe consists in 4,300 women, who constitute the historical average deliveries during the semester in the city of Granada (Spain). The sample collection will be made in medical office's pregnancy control in Granada's hospitals, in their respective health centers and during the second half of 2015. The sample will be stratified and probabilistic. Peculiarities of pregnant women will be taken into account when calculating the size of the study sample. This sample will be made up of 224 women who comply with the inclusion criteria and that have signed the informed consent.

To achieve the project objectives an organization comprising six theoretical and practical phases enabling the scientific development of the project.

During the first phase, the technical and administrative preparation of the project is constructed. Thereafter, the work is divided into two action areas which encompass the collection and data modeling.

The creation of a biological multi-paradigm computer simulation model of the levels of biomarkers in different months of pregnancy and in the various pathologies of pregnant women can be very effective to know the risks that involve high levels of lipids for the mother and for the baby.

ELIGIBILITY:
Exclusion criteria

* Impossibility to participate in the research.
* Restrictive pulmonary disease.
* Cardiac pathology with hemodynamic repercussion.
* Familiar hyperlipidemia.
* Multiple pregnancies.

Inclusion criteria

• Pregnant women healthy and with risk that want participate in a voluntary way in the research and sign the informed consent.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The universe is composed by 4300 women that constitute the historical average of deliveries during a semester in the city of Granada (Spain). The research is projected over women that attend to the pregnancy control consultation into Granada's hospitals during the second semester of 2015. The sample is probabilistic and stratified. To calculate the size of the sample they were considered the characteristics of pregnant women that to be formed by 224 women that comply with the inclusion criteria and that sign the informed consent.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Triglyceride levels | 18 months
  Begins in the 20 weeks and ended 20 days after delivery. Since the 37 week is taken each 72 hours and then daily when an increase of the values occurs and it's followed until 20 days after delivery.
  Measures during this stage are performed with the reagent disk Piccolo®, using the blood analyzer Piccolo express™. It is designed for using in quantitative determination "in vitro" of the total cholesterol, High Density Lipoproteins and triglycerides in a clinic laboratory.
  The levels of normality have been stablished to the following biomarkers:
  Triglycerides levels: under 150 mg/dl, with a high limit between 155 and 199 mg/dl and higher between 200 and 499 mg/dl. During pregnancy it is recommended to keep it under 300 mg/dl.
prolactin levels | 18 months
  Prolactin: 10- 209 ng/ml.
glucose levels | 18 months
  Gestational diabetes: it is diagnose when in the O'Sullivan test the values are equal or superior to the following: blood sugar 105 mg/dl; 1 hour,190 mg/dl; 2 hours, 165 mg/dl and 3 hours, 145 mg/dl.
cholesterol levels | 18 months
  To determine the values of total cholesterol, HDL, LDL and triglycerides the samples should be taken after 8 or 12 hours without eating.
  The test begins after 10 minutes of transferring the sample to the disk. The levels of normality are:
  Total cholesterol: under 200 mg/dl. LDL cholesterol: 40-60 mg/dl, values under 40 mg/dl indicate a higher risk of cardiovascular disease.
Nutritional evaluation | 3 months
  In the first interview to the pregnant woman and after the sign of the informed consent the medical record is performed. Nutritional evaluation is carry out through a validate survey that was published in 2012 by our research team (González Jiménez et al., 2012).
  Bioelectrical impedance was also performed. In clinical history socio demographics variables personal and familiars were collected and anxiety and depressive test were performed (Snaith & Zigmond, 1983).
Collection of samples: mother's milk | 6 months
  It is about to follow the evolution of the process of lactation and the quality of mother's milk. In each group of study three samples are collected: colostrum (2 to 6 days after delivery); transition milk (7 to 21 days after delivery) and maturing milk (after 21 days of delivery).
  Lactogenesis is the process that begins with milk secretion. It is stablished between 24 hours and the sixth day after delivery and is a consequence of the action of prolactin and the low estrogenic level. Before delivery, PRL levels increase but the estrogens of placenta blocked the secretion of glands. The maintaining of lactation requires a continuous suction of the nipple. The estrogenic fall after delivery allows unblock or mammary tissue.

SECONDARY OUTCOMES:
Mother's milk: short-chain fatty acid | 6 months
  According technique developed by the Research Department of Nutrition and Food Science (Journal of Chemistry.2014 ) by gas chromatography using a Perkin Elmer Autosystem gas chromatograph ( Perkin -Elmer , Norwalk , CT , USA ) , equipped with a detector flame ionization (FID ) and a capillary column Supelco 2380 TVSS (30 m × 0.25 mm id , 0.2 um film thickness) .
Mother's milk: Total fatty acid profile | 6 months
  Mass spectrometry using low resolution [ MSP ] with triple quadrupole analyzer (triple -quad ) WATERS model QUATTRO and micro GC Gas Chromatograph model 7890A AGILET , with injectors split / splitless and PTV for capillary columns . Servicos Central Scientific Instrumentation of the UGR ( http://cic.ugr.es/ )
Bioactive peptides | 6 months
  For purification of the peptides the whey are subjected to ion exchange using Dowex 50WX2 resin in the column ( 2.6 x 10 cm , H + -form , 200-400 mesh , Serva , Heidelberg , Germany) according to the procedure described by Farvin et al., 2010 .

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No